CLINICAL TRIAL: NCT07265245
Title: Analogies As A Possible Effective Consultation Tool In Type II Diabetes Mellitus Patients on Insulin: A Retrospective Cohort Study
Brief Title: Evaluating an Analogy-Based Consultation Approach for Insulin-Treated Type 2 Diabetes Patients
Acronym: ANALOGIES01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Muhammad Hanif Bin Omar, Principal Investigator, Ministry of Health, Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NMRR ID-24-00725-QIL
Record Dates: First submitted 2025-11-22; First posted 2025-12-04 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; analogies; M2-PRIME; Consultation module
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- M2-PRIME applied (Experimental): M2-PRIME
  Interventions: Behavioral: M2-PRIME

INTERVENTIONS:
Behavioral: M2-PRIME — Participants received consultations delivered using the M2-PRIME framework, which applies analogy-based education (e.g., the "Garbage and Lorry" model) to improve understanding of diabetes and insulin use.

SUMMARY:
The goal of this retrospective interventional study is to learn whether a new consultation approach called M2-PRIME can help improve blood sugar control in people with type 2 diabetes who use insulin and have high blood sugar levels (HbA1c more than 8.5%).

The main questions are:

1. Does using M2-PRIME during consultations help lower HbA1c (3-month average blood sugar level)?
2. Does using M2-PRIME help lower fasting blood sugar (FBS, morning blood sugar)?

In this study, participants received their regular diabetes care at the Self-Monitoring of Blood Glucose (SMBG) clinic, which runs once a week. Two primary healthcare providers (PHPs) trained in the M2-PRIME framework provided the consultations.

During each visit, PHPs used M2-PRIME to:

1. Build rapport and review the participant's health and lifestyle,
2. Give simple advice about food, activity, and insulin use,
3. Use the "Garbage and Lorry" analogy to explain how the body handles sugar, 4. Educate regarding insulin self-adjustment and monitoring

5. Adjust insulin doses when needed

Each participant had three consultations over six months. Their HbA1c and fasting blood glucose were measured at the start and after six months to see if their blood sugar control improved.

DETAILED DESCRIPTION:
This study is designed to evaluate the effectiveness of a novel analogy-based consultation framework, called M2-PRIME (The Metaphoric Medicine Practical Roadmap for Insulin Management Essentials ), in improving glycaemic control among insulin-treated type 2 diabetes mellitus (T2DM) patients.

The M2-PRIME framework aims to simplify complex diabetes concepts using metaphors and analogies. Its core analogy, the "Garbage and Lorry" model, describes blood sugar as "garbage" that accumulates in the bloodstream, while insulin acts as a "lorry" that carries the sugar into the body's cells, represented as the "factory." The framework is intended to improve understanding, adherence, and motivation among people with T2DM through simplified and unified communication.

This will be a retrospective, single-group pre-post interventional study conducted at a government primary care Self-Monitoring of Blood Glucose (SMBG) clinic in Klinik Kesihatan Senawang, Negeri Sembilan, Malaysia. The clinic runs once a week and is managed by two trained primary healthcare providers (PHPs).

Participants will include adults with insulin-treated T2DM and poor glycaemic control (HbA1c > 8.5%). All participants will have received standard diabetes care at the SMBG clinic, with M2-PRIME introduced as part of routine service improvement. Each participant will have received up to three structured M2-PRIME consultations over six months. Each consultation will include:

1. Building rapport and reviewing medical and lifestyle history,
2. Providing tailored education on diet, physical activity, and medication adherence,
3. Using the "Garbage and Lorry" analogy to explain how insulin helps lower blood sugar
4. Adjusting insulin doses and problem-solving based on self-monitoring results.

The primary outcomes will be changes in HbA1c (%) and fasting blood sugar (FBS, mmol/L) between baseline and six months after the final consultation. Outcome data will be collected from participants who completed follow-up, and will be analyzed using paired-samples statistical tests.

This study has received approval from the Medical Research and Ethics Committee (MREC), Ministry of Health Malaysia (NMRR ID-: 24-00725-QIL, Ref: 24-00725-QIL). Because it involves retrospective analysis of anonymized clinical data from patients who had already received standard care, the requirement for individual informed consent has been waived in accordance with the Declaration of Helsinki (2013) and Malaysian Good Clinical Practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Established T2DM patients, already on insulin therapy regardless of the type of insulin or regime or duration of treatment
* HbA1c at referral more than 8.5%
* Already seen by diabetic educator or dietician prior to referral

Exclusion Criteria:

* Pregnant or found to be pregnant during follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2025-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMAD HANIF B OMAR, MICGP, Principal Investigator — Ministry of Health, Malaysia
Locations (1):
- Klinik Kesihatan Senawang, Seremban, Negeri Sembilan, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
The data and materials necessary to reproduce the findings that includes all of the individual participant data collected during the trial, after de-identification, Study Protocol, Statistical Analysis Plan, Clinical, Study Report, Analytic Code will be made available immediately following publication with no end date. Anyone can access the data, and the data can be used for any purpose. Data are available indefinitely at Open Science Framework https://osf.io/v26ku/overview
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: immediately
Access Criteria: Anyone can access the data, and the data can be used for any purpose
URL: https://osf.io/v26ku/overview

REFERENCES:
- See also: Data Reposition — http://osf.io/v26ku/overview
- Available data/document: IPD Approval letter: MREC APPROVAL LETTER — https://osf.io/v26ku/files/yskbz

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were identified through routine referrals to the Self-Monitoring of Blood Glucose (SMBG) clinic at Klinik Kesihatan Senawang. All eligible adults with insulin-treated type 2 diabetes mellitus and HbA1c greater than 8.5% during the study period were enrolled as part of standard clinical care.
Pre-assignment Details: This study involved a retrospective review of anonymized clinical records of patients who had already received standard care under the SMBG clinic. No randomization or allocation to study groups occurred. The M2-PRIME consultation framework was implemented as part of routine service improvement prior to data extraction. Participants were included in the analysis if they completed at least three consultation sessions with available baseline and follow-up HbA1c data.
Groups:
- M2-PRIME Applied: Participants received routine diabetes care at a primary care Self-Monitoring of Blood Glucose (SMBG) clinic, where consultations were delivered using the M2-PRIME (Metaphoric Medicine Practical Roadmap for Insulin Management Essentials) framework. The framework was used as a structured communication and education approach during standard clinical consultations and did not involve experimental treatments or additional procedures beyond usual care.
  These consultations focuses on patient empowerment on self-adjustment of their insulin based on their SMBG. Participants will then be given an intensification protocol as outlined in the M2-PRIME, with a 6 week appointment to review their condition and SMBG. All diet, lifestyle and clinical guidance follow Malaysia's T2DM CPG. The first consultation lasts up to 30 minutes, depending the complexity of the cases.
  On subsequent appointments, the focus shifts to optimizing patient's insulin based on their lifestyle and diet modification, guided by their latest SMBG. Any issues or concerns are addressed during these sessions. These consultation lasts up to 15 minutes.
Period: Overall Study
Arm/Group | M2-PRIME Applied
Started | 106
Completed | 89
Not Completed | 17
Not completed — Lost to Follow-up | 17

BASELINE CHARACTERISTICS:
Arm/Group | M2-PRIME Applied
Number analyzed (Participants) | 89
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.2 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Baseline HbA1c [Mean (Standard Deviation); unit: Percent] — Baseline HbA1c prior to first consultation using M2-PRIME
  Percent | 11.88 (1.84)
Baseline fasting blood glucose [Mean (Standard Deviation); unit: mmol/L] — Baseline Fasting Blood Glucose (FBS) prior to first consultation using M2-PRIME
  mmol/L | 12.54 (6.32)

OUTCOME MEASURES:

1. Secondary Outcome: Fasting Blood Sugar
Description: Fasting Blood Sugar (FBS) (mmol/L) in 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | M2-PRIME Applied
Number analyzed (Participants) | 89
mmol/L | 9.22 (4.89)

2. Primary Outcome: HbA1c
Description: HbA1c (%) at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Percentage (%) of HbA1c
Arm/Group | M2-PRIME Applied
Number analyzed (Participants) | 89
Percentage (%) of HbA1c | 10.31 (2.01)

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, an average of 6 months.
Description: The intervention involved structured educational consultations only. No medication changes beyond routine clinical care were mandated.
Arm/Group | M2-PRIME Applied
All-Cause Mortality (participants affected / at risk) | 0/89
Serious Adverse Events (participants affected / at risk) | 0/89
Other Adverse Events (participants affected / at risk) | 0/89

LIMITATIONS AND CAVEATS:
Firstly, the study design lacks a control group. Secondly, the relatively high loss to follow-up (16.8%) raises the possibility of selection bias. Thirdly, the short 6-month follow-up period limits conclusions about the long-term sustainability of glycaemic control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT07265245/Prot_SAP_000.pdf